CLINICAL TRIAL: NCT03713125
Title: Early Academic Achievement and Intervention Response: Role of Executive Function
Brief Title: Executive Function in Early Childhood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Laura Cutting, Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 181739; 1R37HD095519-01A1 (NIH)
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Reading Disability
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reading Tutoring Intervention (Active Comparator): 20 hours of one-on-one reading tutoring administered over 6 weeks
  Interventions: Behavioral: Reading Tutoring
- Business as Usual (No Intervention): Instruction as usual within schools

INTERVENTIONS:
Behavioral: Reading Tutoring — 20 hours of 1:1 reading tutoring intervention over 6 weeks
  Arms: Reading Tutoring Intervention

SUMMARY:
Despite the fact that a substantial number of school age children struggle with both reading and math acquisition, the brain mechanisms of the overlapping aspects of reading and math skills, thought in part to be linked via executive functions (EF), have not been unpacked. This project will use a longitudinal design, following children from Kindergarten through 1st grade, to understand how the brain networks associated with reading, math, and EF interact to predict academic outcomes and, in those who struggle academically, intervention response.

DETAILED DESCRIPTION:
This longitudinal study will be conducted with 260 Kindergartners, staggered across multiple cohorts, who are followed through 1st grade. There will be three time points of testing for each cohort: fall of Kindergarten, spring of Kindergarten, and in the fall of 1st grade.

After the third testing time point, in the fall of 1st grade, the bottom 1/3 of readers in the sample will be selected to participate in the intervention arm of the study. These students will be randomly placed in one of two arms: business-as-usual, in which children receive no additional instruction; or the reading intervention condition, in which they receive 20 hours of 1:1 reading intervention over 6 weeks. Children in both sub-sample arms are assessed again after tutoring is complete, in the spring of 1st grade.

Neuroimaging through magnetic resonance imaging (MRI) and functional magnetic resonance imaging (fMRI) will occur as part of study participation in conjunction with testing at fall of Kindergarten, fall of 1st grade, and spring of 1st grade time points.

ELIGIBILITY:
Inclusion Criteria:

1. Children in Kindergarten (approximate ages 4-9 years)
2. Native English speakers

Exclusion Criteria:

1. Children not in Kindergarten at time of enrollment;
2. previous diagnosis of Intellectual Disability;
3. known uncorrectable visual impairment;
4. documented hearing impairment greater than or equal to a 25 decibel (dB) loss;
5. medical contraindication to MRI procedures (e.g., metal devices) - excludes from MRI procedures only;
6. known intelligence quotient (IQ) below 70;
7. a pervasive developmental disorder; and
8. any known neurologic pathology, including epilepsy, spina bifida, cerebral palsy, traumatic brain injury, and brain tumors.
9. Comorbid severe psychiatric disorders will also be excluded, as will those who are taking psychotropic medications, with the exception of stimulant medication for Attention Deficit Hyperactivity Disorder (ADHD). Children who meet criteria for ADHD will be eligible as long as they are not taking psychotropic medications, with the exception of stimulant medication for ADHD.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Woodcock Johnson Tests of Achievement, Fourth Edition (WJ-IV) | Baseline, at study entry (Fall of Kindergarten)
  WJ-IV Letter Word Identification, Word Attack, and Passage Comprehension subtests will be administered in order to assess letter and word recognition accuracy, decoding accuracy and reading comprehension. WJ-IV Calculation and Applied Problems will be administered to assess number identification, basic numeracy skills, and math problem solving. To assess whether cognitive and/or neural metrics of executive function and neural metrics of academic achievement predict academic ability at the same time point.
Change in Woodcock Johnson Tests of Achievement, Fourth Edition (WJ-IV) | Baseline, at study entry (Fall of Kindergarten); and approximately 1 year after baseline (Fall of 1st Grade)
  Change from baseline in reading (as measured by WJ-IV Letter Word Identification, Word Attack, and Passage Comprehension subtests) and math (as measured by WJ-IV Calculation and Applied Problems subtests).
Change in Woodcock Johnson Tests of Achievement, Fourth Edition (WJ-IV) | Approximately 1 year after baseline (Fall of 1st Grade); and approximately 1 year 3 months after baseline (Spring of 1st Grade)
  Change from pre-intervention testing to post-intervention testing in reading (as measured by WJ-IV Letter Word Identification, Word Attack, and Passage Comprehension subtests) and math (as measured by WJ-IV Calculation and Applied Problems subtests).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie E Cutting, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No